CLINICAL TRIAL: NCT05908370
Title: Accuracy of LeFort I Osteotomy Fixation Using Two Plates Versus Four Plates Patient Specific Osteosynthesis. A Randomized Clinical Trial
Brief Title: Accuracy of LeFort I Osteotomy Fixation Using Two Plates Versus Four Plates Patient Specific Osteosynthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Waleed Hossam Mohamed Sabri Ibrahim, Master Candidate at the Faculty of Oral and Dental Medicine, Future University in Egypt, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: (25)11-2021
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Le Fort; I

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxillary orthognathic surgery using 4 patient specific osteosynthesis (4-Plates) (Experimental)
  Interventions: Procedure: Maxillary orthognathic surgery using 4 patient specific osteosynthesis (4-Plates)
- Maxillary orthognathic surgery using 2 patient specific osteosynthesis (2-Plates) (No Intervention)

INTERVENTIONS:
Procedure: Maxillary orthognathic surgery using 4 patient specific osteosynthesis (4-Plates) — Maxillary orthognathic surgery using 4 patient specific osteosynthesis (4-Plates)
  Arms: Maxillary orthognathic surgery using 4 patient specific osteosynthesis (4-Plates)

SUMMARY:
Virtual Surgical planning (VSP) has significantly improved many aspects of oral and maxillofacial surgery. A very important aspect is surgical accuracy and precise transfer of the surgical plan to the operating theatre and reduction of operative time. Conventional treatment planning for orthognathic surgery, although proven to be reliable, has many drawbacks. Computer guided splintless maxillary orthognathic surgery has been recently performed with predictable outcomes. More than one design of PS osteosynthesis has been used in recent trials. Nevertheless, which design is more superior to the other is a topic yet to be addressed. Either a one-piece fixation device spanning the length of the Le Fort 1 osteotomy or the fixation can be provided by more than one device placed at the load bearing buttresses. The superiority of 4 fixating patients specific plates compared to the other will be determined after evaluating many outcomes including accuracy, intra operative time, post-operative complications.

The goal is to take a step towards determining which design is the best for performing splintless maxillary orthognathic surgery in terms of accuracy and least complications for the correction of prevalent dentofacial deformities.

Beside the evaluation of accuracy, the two different designs will be compared in terms of operative time and post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with dentofacial deformity: skeletal class 2, class 3, vertical maxillary excess, Facial asymmetry.
* Patient seeking definitive maxillary or bimaxillary surgical correction and refusing orthodontic camouflage.
* Patient due to receive a non- segmental Le Fort I osteotomy as part of their orthognathic surgery.
* Patient age at least 18 years
* Highly motivated patients.
* Good oral hygiene.
* Patients willing for follow-up, with an informed consent

Exclusion Criteria:

* Medically compromised patients redeeming unfit for general anesthesia
* Pregnancy
* patient had a known allergy to titanium
* Patients with any diseases that may compromise bone or soft tissue healing.
* Patients with local pathosis that may interfere with the bone healing.
* Patient with previous maxillary surgery having hardware that may compromise accuracy of the virtual planning

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Accuracy | 1 week
  Primary outcome will be the positional accuracy of the repositioned maxilla which will be measured via CT scan by superimposing the postoperative maxillary segment obtained from a 1-week postoperative CT with the planned one and the difference is calculated in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Future Univerisity in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided